CLINICAL TRIAL: NCT02894853
Title: Lung Cancer Early Molecular Assessment Trial
Acronym: LEMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); Roche Pharma AG (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: M15LEM; NL54778.031.15 (Other: METC-AVL)
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fluid Therapy; Blood Specimen Collection; Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — both tissue and blood samples will be used
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Liquid (blood) biopsies and tumor biopsy (optional) — Liquid (blood) biopsies: 40 ml (maximal 10 times per patient) Tumor biopsy (optional)

SUMMARY:
The investigators hypothesize that an early molecular profiling, that includes both tissue and blood-bases analysis, for all NSCLC patients, including stage I-III, will increase diagnostic efficiency. When molecular profiles are available at an earlier stage of disease, more patients will benefit from personalized therapy once needed. This will result in both a better quality of life and outcome.

DETAILED DESCRIPTION:
In this prospective multicentre trial tumours of all patients presenting with NSCLC will be profiled upfront, irrespective of disease stage and pathology using both tissue and blood-based genetic testing. A minimal molecular profiling is depicted but other targets will be included in due time. The study is divided in two parts. In the first part participating centres will have a run-in period of half a year in which molecular profiling is performed as is currently standard of care. This period will be used to measure the impact of increased awareness on the diagnostic process. During the second part of the study a comprehensive upfront profiling according to local standards will take place for all NSCLC patients. Liquid (blood) biopsies will be included in order to increase the diagnostic yield for those patients where tissue biopsies are not adequate. Patients will be treated according to standard of care, or included in clinical studies where appropriate. Re-biopsies (both tissue and liquid) will be advocated at the time of establishing disease progression/disseminated disease, and personalized therapy will be initiated according to the existing data from the molecular profiling.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of lung carcinoma or established NSCLC but awaiting start of definitive treatment
* Written informed consent to undergo diagnostic procedure and molecular analysis of the disease.

Exclusion Criteria:

* Not motivated to receive any treatment at any point in time. Patients who consider undergoing treatment in the future are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with NSCLC will be profiled upfront, irrespective of disease stage and pathology using both tissue and blood-based genetic testing
Sampling Method: Non-Probability Sample
Enrollment: 1297 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with EGFR mutation or ALK translocation using the combined tumour tissue and liquid biopsy analysis | 3 years
  Patients with EGFR mutation or ALK translocation using the combined tumour tissue and liquid biopsy analysis

SECONDARY OUTCOMES:
Include the test performance of both techniques in different stage of disease | 3 years
  Test performance of both techniques in different stage of disease
The percentage of patients with a predefined actionable genetic alteration | 3 years
  Patients with a predefined actionable genetic alteration
The costs | 3 years
  The costs
The influence of the liquid biopsies on the diagnostic yield of tissue molecular and pathological analysis. | 3 years
  Liquid biopsies on the diagnostic yield of tissue molecular

CONTACTS AND LOCATIONS:
Overall Officials: Michel van den Heuvel, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuurbiers M, Huang Z, Saelee S, Javey M, de Visser L, van den Broek D, Heuvel MVD, Lovejoy AF, Monkhorst K, Klass D. Biological and technical factors in the assessment of blood-based tumor mutational burden (bTMB) in patients with NSCLC. J Immunother Cancer. 2022 Feb;10(2):e004064. doi: 10.1136/jitc-2021-004064. PMID 35217576